CLINICAL TRIAL: NCT01718899
Title: A Phase 1/2a Dose Escalation Study of PVX-410, a Multi-Peptide Cancer Vaccine, in Patients With Smoldering Multiple Myeloma
Brief Title: Phase 1/2a Study of Cancer Vaccine to Treat Smoldering Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoPep, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-001
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Smoldering Multiple Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma | interventions — PVX-410 vaccine; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PVX-410, .4 mg dose (Experimental): Approximately 3 patients will receive 6, bi-weekly, subcutaneous injections of a .4 mg dose of PVX-410 in combination with an intramuscular injection of Hiltonol (poly ICLC). Patients will complete a 12 week treatment phase and then will be followed for safety, immunogenicity and clinical response for 12 months.
  Interventions: Biological: PVX-410
- PVX-410, .8 mg dose (Experimental): Approximately 10 patients will receive 6, bi-weekly, subcutaneous injections of an .8 mg dose of PVX-410 in combination with an intramuscular injection of Hiltonol (Poly ICLC). Patients will complete a 12 week treatment phase and then will be followed for safety, immunogenicity and clinical response for 12 months.
  Interventions: Biological: PVX-410
- PVX-410 plus lenalidomide (Experimental): Approximately 10 patients will receive 6, bi-weekly, subcutaneous injections of an .8 mg dose of PVX-410 in combination with an intramuscular injection of Hiltonol (Poly ICLC). Patients will also receive 3 cycles of lenalidomide. Patients will complete a 12 week treatment phase and then will be followed for safety, immunogenicity and clinical response for 12 months
  Interventions: Biological: PVX-410

INTERVENTIONS:
Biological: PVX-410 — Approximately 10 patients will receive 6, bi-weekly, subcutaneous injections of a dose of PVX-410 in combination with an intramuscular injection of Hiltonol (Poly ICLC). Patients will complete a 12 week treatment phase and then will be followed for safety, immunogenicity and clinical response for 12 months
  Other Names: Revlimid

SUMMARY:
The purpose of this study is to determine the safety and tolerability of PVX-410, (a cancer vaccine), treatment regimen for patients with smoldering multiple myeloma as a single agent and in combination with lenalidomide.

DETAILED DESCRIPTION:
This is a dose escalation, phase 1/2a study to assess the safety and tolerability of PVX-410, (a multi-peptide cancer vaccine), treatment regimen in patients with smoldering multiple myeloma as a single agent and in combination with lenalidomide.. Approximately 22 patients will receive six (6) bi-weekly, subcutaneous injections of PVX-410 for a total of twelve (12) weeks of treatment. Safety will be monitored throughout the study. Tolerability, immunogenicity and clinical response will also be measured as described in the protocol.

ELIGIBILITY:
* Patient has confirmed clinical diagnosis of SMM according to a definition derived from the International Myeloma Working Group (IMWG) definition: serum M-protein ≥3 g/dL or bone marrow clonal plasma cells (BMPC) greater than or equal to 10%, or both, along with normal organ and marrow function (CRAB) within 4 weeks before baseline.
* C: Absence of hypercalcemia, evidenced by a calcium <10.5 mg/dL.
* R: Absence of renal failure, evidenced by a creatinine <2.0 mg/dL or calculated creatinine clearance (using the Modification of Diet in Renal Disease [MDRD] formula) >50 mL/min.
* A: Absence of anemia, evidenced by a hemoglobin >10 g/dL.
* B: Absence of lytic bone lesions on standard skeletal survey.
* Patient is at higher than average risk of progression to active MM, defined as having 2 or more of the following features:
* Serum monoclonal (M)-protein ≥3 g/dL.
* BMPC greater than or equal to 10%.
* Abnormal serum free light chain (FLC) ratio (0.26-1.65).
* Patient has a life expectancy of greater than 6 months
* Patient is human leukocyte antigen (HLA)-A2 positive.
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Patient has adequate bone marrow function, evidenced by a platelet count ≥75×109/L and an absolute neutrophil count (ANC) ≥1.0×109/L within 2 weeks before baseline.
* Patient has adequate hepatic function, evidenced by a bilirubin ≤2.0 mg/dL and an alanine transaminase (ALT), and aspartate transaminase (AST) ≤2.5× the upper limit of normal (ULN) within 2 weeks before baseline.
* If of child-bearing potential, patient agrees to use adequate birth control measures during study participation.
* If a female of child-bearing potential, patient has negative urine pregnancy test results within 2 weeks before baseline and is not lactating.
* Patient (or his or her legally accepted representative) has provided written informed consent to participate in the study.

Exclusion Criteria:

* Patient has symptomatic multiple myeloma, as defined by any of the following:
* Lytic lesions or pathologic fractures.
* Anemia (hemoglobin <10 g/dL).
* Hypercalcemia (corrected serum calcium >11.5 mg/dL).
* Renal insufficiency (creatinine >2 mg/dL).
* Other: symptomatic hyperviscosity, amyloidosis.
* Patient has abnormal cardiac status, evidenced by any of the following:
* New York Heart Association (NYHA) stage III or IV congestive heart failure (CHF).
* Myocardial infarction within the previous 6 months.
* Symptomatic cardiac arrhythmia requiring treatment or persisting despite treatment.
* Patient is receiving any other investigational agent.
* Patient has a current active infectious disease or positive serology for human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV).
* Patient has a history of or current auto-immune disease.
* Patient has been vaccinated with live attenuated vaccines within 4 weeks before study vaccination.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-11; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
All adverse events will be recorded. | Throughout treatment phase (3 months) and follow up period (12 months)

SECONDARY OUTCOMES:
Immune response to the vaccine will be measured | Designated timepoints during the treatment phase (3 months) and follow up phase (12 months)
  Patient blood samples will be measured for immune response through ELISPOT and Pentamer assays.

OTHER OUTCOMES:
Clinical Response will be measured. | Designated timepoints during the treatment phase (3 months) and follow up phase (12 months)
  Clinical response will be determined by the treating physician according to the International Myeloma Working Group Disease Response Criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Noopur Raje, MD, Principal Investigator — Massachusetts General Hospital; Michael Wang, MD, Principal Investigator — M.D. Anderson Cancer Center; Ajay Nooka, MD, Principal Investigator — Emory University
Locations (6):
- United States (6):
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Illinois Cancer Specialists, Niles, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Texas, MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Nooka AK, Wang ML, Yee AJ, Kaufman JL, Bae J, Peterkin D, Richardson PG, Raje NS. Assessment of Safety and Immunogenicity of PVX-410 Vaccine With or Without Lenalidomide in Patients With Smoldering Multiple Myeloma: A Nonrandomized Clinical Trial. JAMA Oncol. 2018 Dec 1;4(12):e183267. doi: 10.1001/jamaoncol.2018.3267. Epub 2018 Dec 13. PMID 30128502